CLINICAL TRIAL: NCT03980002
Title: A Prospective Multicenter Phase 2 Study of FCR/BR Alternating With Ibrutinib in Treatment-naive Patients With Chronic Lymphocytic Leukemia
Brief Title: A Prospective Multicenter Phase 2 Study of FCR/BR Alternating With Ibrutinib in Treatment-naive Patients With CLL
Acronym: BDHCLL001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, TingyuWang, Attending doctor, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IHBDH-IIT2018009
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Therapeutics; ibrutinib; fludarabine; rituximab; bendamustine; cyclophosphamide; treatment-naive
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Receptors, Fc; ibrutinib; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FCR/BR alternating with ibrutinib (Experimental): FCR/BR→ ibrutinib✖️3months→FCR/BR→ ibrutinib✖️3months→FCR/BR→Maintenance therapy
  Interventions: Drug: FCR and Ibrutinib; Drug: BR and Ibrutinib; Drug: Ibrutinib and Thalidomide

INTERVENTIONS:
Drug: FCR and Ibrutinib — Induction treatment:
  Patients <65 y and without significant comorbidities are given FCR 1or 2 courses (If patients' white blood cell count <10×10^9/L after first course, the second course can be saved). Then, patients takes ibrutinib orally for 3 months alternating with FCR in 2 cylcles.
  1. FCR： F（Fludarabine）：25mg/m2·d，d1-3； C（Cyclophosphamide）：CTX 250mg /m2·d，d1-3； R（Rituximab）：375mg/m2 d0（first course），500mg/m2 d0（subsequent courses）；
  2. Ibrutinib:420mg/d
Drug: BR and Ibrutinib — Induction treatment:
  Patients ≥65y and ≤75 y or <65 y but with comorbidities, are given BR 1or 2 courses (If patients' white blood cell count drop to below10×10^9/Lafter first course, the second course can be saved). Then, patients takes ibrutinib orally for 3 months alternating with BR in 2 cylcles. 1.BR： B（Bendamustine）：90mg/m2·d，d1-2； R（Rituximab）：375mg/m2 d0（first course），500mg/m2 d0（subsequent courses）； 2. Ibrutinib: 420mg/d
Drug: Ibrutinib and Thalidomide — Maintenance treatment:
  After induction treatment, recommend ( but not mandatory) Ibrutinib or thalidomide monotherapy(according to patients preferrance) for MRD-positive patients.For MRD-negative patients, recommend ( but not mandatory) no maintenance therapy.

SUMMARY:
This is a prospective multicenter phase 2 study designed with the purpose to evaluate the response rate and safety of treatment with FCR/BR alternating with ibrutinib in treatment-naive patients with chronic lymphocytic leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 years and ≤ 75 of age.
2. Diagnosis of CLL/SLL that meets IWCLL diagnostic criteria.
3. Treatment-naive patients. Those patients received short-term substandard treatment are permitted if meet all the items listed below:

   1. Untreated with combined chemotherapy such as CHOP ,COP and so on.
   2. Unteated with chemotherapy regimens including fludarabine and bendamustine.
   3. Unteated with Ibrutinib.
   4. If treated with chlorambucil or cyclophosphamide,should less than 3 weeks.
   5. If treated with interferon, should less than 6 months.
   6. No objective response are achieved (PR or CR).
4. CLL/SLL requiring treatment as defined by at least one of the following criteria:

   1. Development of, or worsening of, anemia to Hb<100g/L (non-hemolytic) .
   2. Development of, or worsening of, thrombocytopenia to PLT<100,000/L.
   3. Massive (≥ 6 cm below left costal margin), progressive or symptomatic splenomegaly.
   4. Massive nodes (≥ 10 cm in longest diameter), or progressive or symptomatic lymphadenopathy .
   5. Progressive lymphocytosis with an increase of > 50% over a 2-month period or lymphocyte-doubling time of < 6 months. Lymphocyte-doubling time may be obtained by linear regression extrapolation of absolute lymphocyte counts obtained at intervals of 2 weeks over an observation period of 2 to 3 months. In patients with initial blood lymphocyte counts of < 30,000/L, LDT should not be used as a single parameter to define treatment indication. In addition, factors contributing to lymphocytosis or lymphadenopathy other than CLL/SLL (eg, infection, use glucocorticoid) should be excluded. f)Symptomatic or functional extranodal sites involved s (eg. Skin,kidney, lungs and so on).

   g)Constitutional symptoms, defined as any 1 or more of the following disease-related symptoms or signs: i. Unintentional weight loss of ≥ 10% within the previous 6 months ii.Significant fatigue (ie, inability to work or perform usual activities)
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
6. Expected to survival period for 3 months or more.

Exclusion Criteria:

1. History of malignant tumour except CLL in the past 1year(including active central nervous system (CNS) involvement with lymphoma).
2. Transformed to large cell lymphoma manifested by clinical evidence, or progressed to prolymphocytic leukemia(PLL).
3. Have active autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura, and require treatment.
4. Inadequate hepatic and renal function defined as: AST and ALT >4.0 x upper limit of normal (ULN), bilirubin >2.0 x upper limit of normal (ULN), Adequate renal function defined by serum creatinine >1.5 x upper limit of normal (ULN),unrelated to lymphoma.
5. Severe or uncontrolled infection.
6. Central nervous system (CNS) dysfunction with clinical manifestation.
7. Other serious medical diseases that may affect the study（eg. Uncontrolled diabetes, gastric ulcer, other severe cardiopulmonary disease),and final decided by the investigator.
8. Ongoing and uncontrolled bleeding
9. History of major life-threatening bleeding, especially due to irreversible cause.
10. Requirement for continuous anticoagulation drugs.
11. Major surgery within 30 days(excluding lymph node biopsy).
12. Pregnant or Lactating women, or women of reproductive age refusal to take contraceptive measures.
13. Allergy to any drug used in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
CRR | 3 months after completion of induction therapy
  Rate of complete remission

SECONDARY OUTCOMES:
ORR | 3 months after completion of induction therapy
  Overall Response Rate
OS | 5 years
  Overall survival
PFS | 5 years
  Progression-free survival
MRD negative rate | 3 months after completion of induction therapy
  the rate of undetectable tumor cells in bone marrow and/or peripheral blood by multicolor flow cytometry
DoR | 5 years
  Duration of Response
Treatment-related side effects | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Zengjun Li, Principal Investigator — Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang T, Yan Y, Wang H, Sun Y, Liu X, Lyu R, Xiong W, An G, Liu W, Xu Y, Deng S, Wang Q, Du C, Huang L, Zou D, Zhao Y, Qiu L, Li Z, Yi S. Ibrutinib alternating with three cycles of interval fludarabine, cyclophosphamide, and rituximab (FCR) in adults with untreated chronic lymphocytic leukaemia as time-limited regimen: a single-arm, multicentre phase 2 trial in China. EClinicalMedicine. 2025 Dec 5;90:103688. doi: 10.1016/j.eclinm.2025.103688. eCollection 2025 Dec. PMID 41497516